CLINICAL TRIAL: NCT03123809
Title: Combined Gastric Electrical Stimulation (GES) and Pyloroplasty for the Treatment of Gastroparesis: Can Pyloroplasty be Effective Without GES?
Brief Title: Gastric Electrical Stimulation (GES) and Pyloroplasty for the Treatment of Gastroparesis
Acronym: GES+PP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Irene Sarosiek, Professor of Medicine, Texas Tech University Health Sciences Center, El Paso
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E16156
Record Dates: First submitted 2017-04-13; First posted 2017-04-21 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Gastroparesis
Keywords: Diabetes Mellitus; gastroparesis; gastric electrical stimulation; pyloroplasty; Idiopathic -unknown etiology
MeSH Terms: conditions — Gastroparesis; Diabetes Mellitus | interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: Based on confidential code set up for this study, there will be a randomized assigment for patients to have their GES devices turn ON or OFF. Half of these patients will be in each arm.
Who Masked: Participant, Investigator
Masking Description: Patient and clinical investigators are going to be blinded in regards to the status of GES (if it is ON or OFF) for 3 months after surgery. One non-clinical investigator is assigned to serve as un-blind person , who is going to generate a master list of participants by dividing them into two groups based on their etiologies (diabetic or idiopathic). All effort would be to include similar numbers of idiopathic and diabetic patients in each intervention group based on a block randomization method, allowing for GES to be turned ON at the surgery, or it will stay OFF for the 3 month during the blind portion of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (2):
- Gastric Electrical Stimulation (GES) ON (Active Comparator): Gastric Electrical Stimulation (GES) system involves surgical implantation of a pulse generator in the abdominal wall and 2 electrodes into the muscularis propria of the stomach.
  After surgery this group of GP patients will have their GES programed and system will be turned ON for 3 months during a double-blind phase of the study. This step will be followed with additional 3 months of active stimulation (GES System will be turned ON) as it is described in the protocol.Therefore all subjects in this arm will receive overall 6 months of intervention, which will be provided by the active stimulation of GES System (GES turned ON for 6 months).
  Interventions: Device: Gastric Electrical Stimulation (GES) System
- Gastric Electrical Stimulation (GES) OFF (Placebo Comparator): Gastric Electrical Stimulation (GES) system involves surgical implantation of a pulse generator in the abdominal wall and 2 electrodes into the muscularis propria of the stomach.
  After surgery this group of GP patients will have their GES programed and system will be turned OFF for 3 months.This step will be followed with additional 3 months of active stimulation (GES System will be turned ON) as it is described in the protocol. Therefore all subjects in this arm will receive first 3 months of non GES intervention (GES System OFF), and 3 following months of active intervention which will be provided by the stimulation of GES System (GES turned ON for 3 months).
  Interventions: Device: Gastric Electrical Stimulation (GES) System

INTERVENTIONS:
Device: Gastric Electrical Stimulation (GES) System — Implantable GES System will be turned ON as an active intervention providing electrical stimulation to the muscle of stomach for 6 months in patients from the first arm, versus 3 months only of active stimulation in patients who are randomized to be in the second arm of the study. GES works by utilizing following parameters: Current 5 mA; Pulse Width 330µsec; Rate 14 Hz; Time ON 0.1 sec; Time OFF 5.0 sec.
  Other Names: Enterra II Therapy System INS Model 37800;

SUMMARY:
Gastroparesis (GP) is describing a condition when stomach does not empty as fast as it should. This fact creates the situation, when food stays in the stomach for a long time and it causes symptoms of nausea, vomiting, loss of appetite, bloating, inability to finish normal size meal and abdominal pain. There are not many drugs available to treat this condition and majority of gastroparetic patients are not responding well to them after they are on it for some time. Many investigators are able to implant Gastric Stimulator System (GES) under FDA approved status of Humanitarian Device Exemption (HDE) definition. In the last few years it became possible to add another surgical procedure, which is called pyloroplasty (making bigger opening on the end of stomach), may help even more as it is also increasing the rate of the emptying of the stomach. Therefore this study is proposing to evaluate if GES in combination with pyloroplasty is much better than pyloroplasty alone. For this reason, two of these procedures will be introduced surgically at the same time, but GES devices will not be turn ON in half of these participants for 3 months. After that time all subjects will have their devices turned ON. All subjects will be asked to evaluate their symptoms of gastroparesis and their quality of life during clinical visits, and investigators will conduct pathological analyses of tissue obtained during surgery.

DETAILED DESCRIPTION:
GES system (Enterra Therapy) involves surgical implantation of a pulse generator in the abdominal wall and 2 electrodes into the muscularis propria of the stomach. Well established procedure, called pyloroplasty, will be performed during the implantation of GES system, therefore all participants will have both surgeries done at the same time. Half of them will be randomized to keep GES ON after surgery, and other half will have GES turned OFF for 3 months.

Both groups will be followed for additional 3 more months. Study related questionnaires and diagnostic/ clinical tests will be obtained at all points of interest of this study.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of GP for > 1 year and refractoriness to anti-emetics and prokinetics; more than 7 emetic episodes per week;
* Delayed GE (gastric retention greater than 60% at 2 h and/or greater than 10% at 4 h) based on a 4-h standardized radionuclide solid meal test

Exclusion Criteria:

* Organic or pseudo-obstruction, primary eating or swallowing disorders, positive pregnancy test result, psychogenic vomiting, peritoneal dialysis, drug dependent, morbid obesity, active malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Changes of total gastroparesis symptom scores (TSS) | up to 7 months
  Severity and frequency of gastroparesis symptoms will be assess at baseline /surgery, after 3 months of randomized phase (GES ON or OFF), and at the end of 3 months of clinical follow up visit.

SECONDARY OUTCOMES:
Total Symptom Score (TSS) with severity and frequency of gastroparesis symptoms in each etiological subgroup of patients | Up to 7 months
  TSS in diabetic and idiopathic sub-group of gastroparetic patients will be compared and analyzed (if adequate number of patients will be in each subgroup)
Associations between changes in gastric emptying and TSS | Up to 7 months
  Statistical analyses of any possible correlation between retention of GET study meal and gastroparesis symptoms will be asses at the end of randomized phase of the study.
Percentage of changes of gastric emptying retention of the radiolabeled meal (%) at 2-4 hrs | up to 7 months
  Scintigraphy Gastric Emptying Test (GET) will be recorded at baseline and after 3 months of randomized phase (GES ON or OFF)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Sarosiek, MD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Sciences Center, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarosiek I, Bashashati M, Davis BR, Espino K, Vasquez D, Torelli R, Bright T, Sarosiek J, Diaz JR, Padilla O, Dwivedi AK, McCallum RW. Combined Gastric Electrical Stimulation and Pyloroplasty in Gastroparesis: A Randomized Clinical Trial. JAMA Netw Open. 2025 Dec 1;8(12):e2546332. doi: 10.1001/jamanetworkopen.2025.46332. PMID 41364437